CLINICAL TRIAL: NCT07163494
Title: Assessment of Occlusal Sensitivity to Articulating Foils in Patients With Temporomandibular Disorders Compared to Healthy Controls: A Case-Control Study
Brief Title: Occlusal Sensitivity to Articulating Foils in Patients With Temporomandibular Disorders and Healthy Controls
Acronym: SENFOIL
Status: Not yet recruiting | Type: Observational
Sponsor: University of Zagreb (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Marko Zlendić, DMD, PhD, Assistant, University of Zagreb
Other Study IDs: 05-PA-30-22-11/2023; SFZG-07-2025_LIPOR (Other Grant/Funding Number: Croation National Recovery and Resilience Plan)
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Disorder (TMD); Chronic Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group
- control group

SUMMARY:
Occlusal sensitivity refers to the ability to detect fine objects placed between opposing teeth during biting or in maximum intercuspation. Two main approaches are commonly used to assess occlusal sensitivity and the periodontal sensory threshold: one measures the minimal detectable force using monofilaments, while the other evaluates the sensitivity threshold to interocclusal thickness with articulating foils. In healthy individuals, occlusal sensitivity ranges from 2 µm to 77 µm (average 24 µm) and tends to decrease with age. Periodontal mechanoreceptors are primarily responsible for this function, although studies indicate that other mechanoreceptors may contribute, especially in individuals with implants or prostheses. Evidence suggests that patients with painful temporomandibular disorders (TMD) may have reduced occlusal sensitivity and show less adaptability to occlusal interferences than healthy subjects. This observational case-control study assesses differences in occlusal sensitivity between patients with pain-related TMD and healthy controls. The study will also explore the relationship between sensory sensitivity, psychosomatic characteristics, and the clinical manifestations of TMD. The TMD group will include patients from the Department of Removable Prosthodontics and the Department of Oral Medicine at the University of Zagreb School of Dental Medicine, diagnosed with pain-related TMD (including myalgia, referred myofascial pain, and/or arthralgia) according to the DC/TMD criteria. The control group will consist of healthy volunteers matched for age and sex, with no neurological alterations in sensory function. The study has been approved by the Ethics Committee of the University of Zagreb School of Dental Medicine and will be conducted in accordance with the Declaration of Helsinki. All participants will receive detailed information about the study and provide written informed consent before participation. The experimental procedure will test occlusal sensitivity by assessing the ability of participants to detect different thicknesses of articulating foils, applied in randomised order between upper and lower molars, including a sham test. Participants will report whether they detect the foil, and their responses will be recorded for subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Reported pain in the temporomandibular joint (TMJ) and/or masticatory muscles persists for more than 3 months.

Spontaneous pain >30 mm on the Visual Analogue Scale (VAS) at the time of the first examination.

-

Exclusion Criteria:

Loss of posterior teeth leads to loss of occlusal support zones.

Posterior removable dentures.

Poor oral hygiene or periodontal disease.

Orofacial pathology unrelated to TMD diagnosis.

Acute pain (duration <3 months).

History of head and neck trauma.

Headache not related to TMD (according to the International Classification of Headache Disorders, ICHD-II).

Pain caused by fibromyalgia.

Systemic diseases or diagnosed psychiatric disorders.

History of pain medication abuse or current substance abuse.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants will be Caucasian, of Middle or Southern European descent. The study will include employees of the Department of Dental Medicine at the Clinical Hospital Centre Zagreb, as well as employees and students of the University of Zagreb School of Dental Medicine, along with healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Occlusal Sensitivity Threshold | Up to 1 hour per participant.
Case-Control Comparison | Up to 1 hour per participant.

SECONDARY OUTCOMES:
Clinical TMD Manifestation and Occlusal Sensitivity | Up to 1 hour per participant.

DOCUMENTS (1):
  • Study Protocol (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07163494/Prot_000.pdf